CLINICAL TRIAL: NCT04841759
Title: The Effects of a Multi-factorial Rehabilitation Program for Healthcare Workers Suffering From Post-COVID-19 Fatigue Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Richard Crevenna, Univ.-Prof. Dr. MBA MMSc, Head of Department of Physical Medicine, Rehabilitation and Occupational Medicine, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1181/2021
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
Keywords: Long-COVID; SARS-CoV fatigue syndrome; Exercise; Rehabilitation
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Stratification regarding post-COVID-19 fatigue syndrome at baseline yes/no
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post COVID-19 fatigue at baseline "yes" (Experimental): SARS-CoV2 survivor who attends the exercise program and suffers from post-COVID-19 fatigue Syndrome according to the Post-Covid-19-Functional Scale (PCFS)
  Interventions: Other: Exercise
- Post COVID-19 fatigue at baseline "no" (Active Comparator): SARS-CoV2 survivor who attends the exercise program and doesn't suffer from post-COVID-19 fatigue Syndrome according to the Post-Covid-19-Functional Scale (PCFS)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 8 week exercise program, nutritional & psychological consultation

SUMMARY:
The SARS-CoV2 pandemic has kept the world in suspense for over a year now. Almost 100 million people around the world have contracted COVID-19 to date and over 2 million people have died of COVID-19 by the end of January 2021.

Despite the tragedy of these deaths, it must be pointed out at this point that the number of COVID-19 survivors is significantly larger. These COVID-19 survivors are now the focus of interest in rehabilitation measures, as it has been shown that survival of the disease does not go hand in hand with a complete cure. Thirty-five percent of all COVID-19 survivors and 87% of the COVID-19 survivors who were hospitalized in the course of their illness suffer from after-effects that are currently summarized as post-COVID fatigue syndrome also known as "Long-COVID".

As health care workers are at higher risk of contracting SARS CoV2 and furthermore, considering their central role in the overcoming of this pandemic, a COVID-19 rehabilitation program for healthcare workers of the Medical University of Vienna, Austria as well as the General Hospital of Vienna, Austria - together the second-largest university-clinic in the world - was developed as part of workplace health promotion. Nowadays, the fatigue syndrome is primarily known as a side effect of cancer treatment and thus from the rehabilitation of cancer patients. Cancer-related fatigue is a massive limiting side effect for patients and the currently most effective treatment strategy against cancer-associated fatigue syndrome is physical training.

The idea for this current project is, that physical exercise might have similar effects on post-SARS-CoV2 fatigue as it has on cancer-related fatigue.

The current study evaluates the effects of this primarily exercise-based rehabilitation program on Long-COVID fatigue.

DETAILED DESCRIPTION:
Employees of the Medical University of Vienna, Austria and the General Hospital of Vienna, Austria who survived a SARS-CoV2 infection will be invited to take part in an eight weeks post-COVID-19 rehabilitation program which is part of a workplace health promotion measure. This program consists of eight weeks of exercising (twice per week supervised resistance training + individual, heart-rate controlled endurance training recommendations) with a sports scientist and a sports medicine specialist, complemented by one session of nutrition consultation with a nutritionist and two sessions of psychological consultation with a clinical psychologist.

Parallel to this workplace health promotion program, the scientific evaluation of this intevention will be undertaken via this study.

ELIGIBILITY:
Inclusion Criteria:

* Employees of the Medical University of Vienna, Austria or the General Hospital of Vienna, Austria
* survived COVID-19 infection

Exclusion Criteria:

* acute COVID-19 infection
* serious, uncontrolled diseases of the cardiovascular system
* insufficient language skills to complete the study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Change of maximum oxygen uptake (VO2max) over time-points (baseline - 4 weeks - 8 weeks) assessed during cardio-pulmonary exercise testing (CPET) | Baseline, 4 weeks, 8 weeks
  Measurement of VO2max during an exhaustive CPET is the gold standard for objectifying cardiopulmonary performance and detecting any cardiovascular risks under stress. VO2max will be measured in ml/kg bodyweight.This examination is the gold standard for objectifying cardiopulmonary performance and detecting any cardiovascular risks under stress.

SECONDARY OUTCOMES:
Change of walking distance during a six minutes walk test (6MWT) over time-points (baseline - 4 weeks - 8 weeks) | Baseline, 4 weeks, 8 weeks
  The 6MWT is used, among other things, to assess and control cardiovascular and pulmonary performance below the anaerobic threshold. This test is used for the clinical evaluation of the basic motor property endurance and measures the distance a patient can walk as quickly as possible on a flat, hard surface in a period of 6 minutes. It will be measured in meters.
Change of numbers over time-points (baseline - 4 weeks - 8 weeks) how often someone can stand up and sit down on a chair within 30 seconds during a 30-seconds sit-to-stand test (30secSTS) | Baseline, 4 weeks, 8 weeks
  The 30seconds Sit-to-Stand test is a well-established functional test used to estimate the strength endurance of the lower extremities and describes how often the test person can get up from a chair and sit down again in a period of 30 seconds. In patients suffering from chronic obstructive pulmonary disease (COPD), the 30seconds sit-to-stand test has proven to be a valid and reliable parameter.
Change of absolute body fat over time-points (baseline - 4 weeks - 8 weeks) via Bioelectrical Impedance Analysis (BiA) | Baseline, 4 weeks, 8 weeks
  BiA is a non-invasive method for measuring body composition and serves as a basis for assessing metabolic disease risks among others by measuring body fat in absolute (kg) numbers.
Change of body fat percentage over time-points (baseline - 4 weeks - 8 weeks) via Bioelectrical Impedance Analysis (BiA) | Baseline, 4 weeks, 8 weeks
  BiA is a non-invasive method for measuring body composition and serves as a basis for assessing metabolic disease risks among others by measuring body fat in relative (%) numbers.
Change of absolute Lean Body Mass (LBM) over time-points (baseline - 4 weeks - 8 weeks) via Bioelectrical Impedance Analysis (BiA) | Baseline, 4 weeks, 8 weeks
  BiA is a non-invasive method for measuring body composition and serves as a basis for assessing metabolic disease risks among others by measuring lean body mass in absolute (kg) numbers.
Change of realtive Lean Body Mass (LBM) over time-points (baseline - 4 weeks - 8 weeks) via Bioelectrical Impedance Analysis (BiA) | Baseline, 4 weeks, 8 weeks
  BiA is a non-invasive method for measuring body composition and serves as a basis for assessing metabolic disease risks among others by measuring lean body mass in relative (%) numbers.
Change of generalized anxiety measured over time-points (baseline - 4 weeks - 8 weeks) via Generalized Anxiety Disorder Scale-7 (GAD-7) | Baseline, 4 weeks, 8 weeks
  The GAD-7 (Generalized Anxiety Disorder 7) is a module of the health questionnaire for patients (PHQ-D), which was designed to identify patients with generalized anxiety disorder and to record the severity of symptoms of generalized anxiety (7 items). Scores range from 0 to 21 points with low scores representing low general anxiety and high scores representing high general anxiety.
Change of depression measured over time-points (baseline - 4 weeks - 8 weeks) via the Patient Health Questionnaire-9 (PHQ-9) | Baseline, 4 weeks, 8 weeks
  The questionnaire PHQ-9 corresponds to the depression module of the health questionnaire for patients (PHQ-D). It was developed as a screening instrument for the diagnosis of depression for routine use in the somatic medical field (9 items). Scores range from 0 to 27 points with low scores representing low levels of depression and high scores representing high levels of depression.
Change of mental stress measured over time-points (baseline - 4 weeks - 8 weeks) via Perceived Stress Scale (PSS-10) | Baseline, 4 weeks, 8 weeks
  The PSS-10 measures the subjective experience of stress. It records the dimensions of self-efficacy and helplessness in two scales, as well as an overall stress score (10 items). Scores range from 0 to 50 points with low scores representing low stress levels and high scores representing high stress levels.
Change of fatigue measured over time-points (baseline - 4 weeks - 8 weeks) via Brief Fatigue Inventory (BFI) | Baseline, 4 weeks, 8 weeks
  The BFI measures the severity and extent of fatigue. The questionnaire covers six dimensions: activity, mood, ability to walk, work, relationship with other people and joie de vivre (10 items). Scores range from 0 to 10 points with low scores representing low fatigue and high scores representing high fatigue.
Change of resilience measured over time-points (baseline - 4 weeks - 8 weeks) via Brief Resilience Scale (BRS) | Baseline, 4 weeks, 8 weeks
  The Brief Resilience Scale measures resilience, the ability to successfully cope with difficult, stressful situations or to recover quickly from them (6 items). Scores range from 1 to 5 points with low scores representing low resilience and high scores representing high resilience.
Change and time kinetics of handgrip strength (HGS) over time-points (baseline and before each exercise session) measured via handgrip Dynamometer. | Baseline, and before every supervised resistance exercise session
  Data on the fist force in kg (measurement of the basic motor property force), which are collected using a JAMAR® dynamometer.
Change and time kinetics of physical and functional limitations of COVID-19 survivors over time-points (baseline and before each exercise session) via Post-Covid-19-Functional Scale (PCFS) | Baseline, and before every supervised resistance exercise session
  The Post-COVID-19 Functional Scale is a questionnaire for self-assessment of physical and functional limitations after a COVID-19 infection. It ranges from 0 (no functional impairment) to 4 (severe functional impairments).
Change of work ability over time-points (baseline, 4 weeks, 8 weeks) via Work Ability Index (WAI) questionnaire. | Baseline, 4 weeks, 8 weeks
  The Work Ability Index (WAI) is a measuring instrument for recording the work ability of employees. The WAI is a questionnaire that is filled out either by the respondents themselves or by third parties, e.g. company doctors during the company medical examination. The WAI is predictive of reintegration into working life after workplace-specific rehabilitation against back pain. WAI scores range from 7-27 (poor), over 28-36 (moderate), and 37 to 43 (good) to 44-49 (very good).
Change of troponin (TnT) over time-points (baseline - 4 weeks - 8 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks
  TnT (0 - 14 ng/L) is a heart-specific and very sensitive marker for myocardial damage in case of elevated values
Change of BNP over time-points (baseline - 4 weeks - 8 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks
  BNP (0 - 125 pg/ml) is increased in cardiac insufficiency and increased volume load on the heart
Change of CK-MB over time-points (baseline - 4 weeks - 8 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks
  CK-MB (< 24 U/l) are elevated in cardiac muscle diseases e.g. myocardial infarction, myocarditis, ischemic conditions e.g. angina pectoris, or for the differential diagnosis of muscle diseases
Change of HS-CRP over time-points (baseline - 4 weeks - 8 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks
  CRP (< 0,5 mg/dl) is an "acute phase protein" which increases in infections (bacterial, less viral and fungi), inflammation, post-OP, malignant processes; ultra-sensitive CRP is additionally a risk assessment marker of aterosclerosis
Change of IL-6 over time-points (baseline - 4 weeks - 8 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks
  IL-6 (<= 7 pg/mL) is a mediator of the immune system and elevated in inflammatory processes
Change of cholesterol over time-points (baseline - 4 weeks - 8 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks
  Cholesterol (< 200 mg/dL) is a risk factor for early atherosclerosis
Change of triglycerides over time-points (baseline - 4 weeks - 8 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks
  Triglycerides (< 150 mg/dl) increased in primary hyperlipidemia as a risk faktor for cardiovascular diseases
Change of distance walked in meters per day over time | From the first exercise session over 8 weeks until the last exercise session (daily)
  Spare time physical activity is a key indicator for physical function and will be measured via activity tracker
Change of time of physical activity per day in minutes over time | From the first exercise session over 8 weeks until the last exercise session (daily)
  Spare time physical activity is a key indicator for physical function and will be measured via activity tracker
Change of step count per day over time | From the first exercise session over 8 weeks until the last exercise session (daily)
  Spare time physical activity is a key indicator for physical function and will be measured via activity tracker
Change of average heart rate per day over time | From the first exercise session over 8 weeks until the last exercise session (daily)
  A low average heart rate during activities of daily living is an indicator for a relatively low cardiovascular load
Change of maximum heart rate per day over time | From the first exercise session over 8 weeks until the last exercise session (daily)
  A low maximum heart rate during activities of daily living is an indicator for a relatively lower level of cardiovascular load
Change of average oxygen saturation (in %) per day over time | From the first exercise session over 8 weeks until the last exercise session (daily)
  A high oxygen saturation is an indicator for a well functioning gas exchange in the lungs and distribution into the circulatory system
Change of Mild Cognitive Impairment over time-points (baseline, 8 weeks) via Montreal Cognitive Assessment (MoCA) | Baseline, 8 weeks
  The MoCA test is a screening instrument for Mild Cognitive Impairment. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
Change of sleep quality over time points (baseline, 4 weeks, 8 weeks) via Insomnia Severity Index (ISI) | Baseline, 4 weeks, 8 weeks
  The Insomnia Severity Index (ISI) is a brief self-report instrument measuring the patient's perception of both nocturnal and diurnal symptoms of insomnia.

OTHER OUTCOMES:
Status of bone resorption at baseline | Baseline only
  Carboxy-terminal type I collagen (CTX-1; 0.003-0.44 ng/ml) is a marker of bone resorption.
Status of bone formation at baseline | Baseline only
  Procollagen type 1 amino-terminal propeptide (P1NP; 20-92 ng/ml) is an early marker of bone formation.
Status of bone turnover at baseline | Baseline only
  Bone-specific alkaline phosphatase (BAP) is used to detect minor changes in bone turnover.
Status of bone mineralization at baseline | Baseline only
  Osteocalcin (Oc; 11-46 ng/ml) is a late marker of bone formation.
Status of calcium metabolism at baseline | Baseline only
  25-OH-vitamin D (75-250 nmol/l) is the precursor for calcitriol, the active form of vitamin D which is essential for calcium metabolism
Status of serum calcium concentration regulation at baseline | Baseline only
  Parathyroid hormone (PTH; 15-65 pg/ml) regulates the serum calcium concentration through its effects on bone, kidney, and intestine.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Tenforde MW, Kim SS, Lindsell CJ, Billig Rose E, Shapiro NI, Files DC, Gibbs KW, Erickson HL, Steingrub JS, Smithline HA, Gong MN, Aboodi MS, Exline MC, Henning DJ, Wilson JG, Khan A, Qadir N, Brown SM, Peltan ID, Rice TW, Hager DN, Ginde AA, Stubblefield WB, Patel MM, Self WH, Feldstein LR; IVY Network Investigators; CDC COVID-19 Response Team; IVY Network Investigators. Symptom Duration and Risk Factors for Delayed Return to Usual Health Among Outpatients with COVID-19 in a Multistate Health Care Systems Network - United States, March-June 2020. MMWR Morb Mortal Wkly Rep. 2020 Jul 31;69(30):993-998. doi: 10.15585/mmwr.mm6930e1. PMID 32730238
- [Background] Belli S, Balbi B, Prince I, Cattaneo D, Masocco F, Zaccaria S, Bertalli L, Cattini F, Lomazzo A, Dal Negro F, Giardini M, Franssen FME, Janssen DJA, Spruit MA. Low physical functioning and impaired performance of activities of daily life in COVID-19 patients who survived hospitalisation. Eur Respir J. 2020 Oct 15;56(4):2002096. doi: 10.1183/13993003.02096-2020. Print 2020 Oct. PMID 32764112
- [Background] Halpin SJ, McIvor C, Whyatt G, Adams A, Harvey O, McLean L, Walshaw C, Kemp S, Corrado J, Singh R, Collins T, O'Connor RJ, Sivan M. Postdischarge symptoms and rehabilitation needs in survivors of COVID-19 infection: A cross-sectional evaluation. J Med Virol. 2021 Feb;93(2):1013-1022. doi: 10.1002/jmv.26368. Epub 2020 Aug 17. PMID 32729939
- [Background] The Lancet. COVID-19: protecting health-care workers. Lancet. 2020 Mar 21;395(10228):922. doi: 10.1016/S0140-6736(20)30644-9. No abstract available. PMID 32199474
- [Background] Barranco R, Ventura F. Covid-19 and infection in health-care workers: An emerging problem. Med Leg J. 2020 Jul;88(2):65-66. doi: 10.1177/0025817220923694. Epub 2020 May 22. PMID 32441196
- [Background] Salazar de Pablo G, Vaquerizo-Serrano J, Catalan A, Arango C, Moreno C, Ferre F, Shin JI, Sullivan S, Brondino N, Solmi M, Fusar-Poli P. Impact of coronavirus syndromes on physical and mental health of health care workers: Systematic review and meta-analysis. J Affect Disord. 2020 Oct 1;275:48-57. doi: 10.1016/j.jad.2020.06.022. Epub 2020 Jun 25. PMID 32658823
- [Background] Hilfiker R, Meichtry A, Eicher M, Nilsson Balfe L, Knols RH, Verra ML, Taeymans J. Exercise and other non-pharmaceutical interventions for cancer-related fatigue in patients during or after cancer treatment: a systematic review incorporating an indirect-comparisons meta-analysis. Br J Sports Med. 2018 May;52(10):651-658. doi: 10.1136/bjsports-2016-096422. Epub 2017 May 13. PMID 28501804
- [Background] Wood LJ, Nail LM, Winters KA. Does muscle-derived interleukin-6 mediate some of the beneficial effects of exercise on cancer treatment-related fatigue? Oncol Nurs Forum. 2009 Sep;36(5):519-24. doi: 10.1188/09.ONF.519-524. PMID 19726392
- [Background] Marzetti E, Calvani R, Tosato M, Cesari M, Di Bari M, Cherubini A, Broccatelli M, Savera G, D'Elia M, Pahor M, Bernabei R, Landi F; SPRINTT Consortium. Physical activity and exercise as countermeasures to physical frailty and sarcopenia. Aging Clin Exp Res. 2017 Feb;29(1):35-42. doi: 10.1007/s40520-016-0705-4. Epub 2017 Feb 8. PMID 28181204
- [Background] Klok FA, Boon GJAM, Barco S, Endres M, Geelhoed JJM, Knauss S, Rezek SA, Spruit MA, Vehreschild J, Siegerink B. The Post-COVID-19 Functional Status scale: a tool to measure functional status over time after COVID-19. Eur Respir J. 2020 Jul 2;56(1):2001494. doi: 10.1183/13993003.01494-2020. Print 2020 Jul. PMID 32398306
- [Derived] Hasenoehrl T, Palma S, Huber DF, Kastl S, Steiner M, Jordakieva G, Crevenna R. Post-COVID: effects of physical exercise on functional status and work ability in health care personnel. Disabil Rehabil. 2023 Sep;45(18):2872-2878. doi: 10.1080/09638288.2022.2111467. Epub 2022 Aug 18. PMID 35980383
- See also: WHO (2021) WHO Coronavirus Disease (COVID-19) — https://covid19.who.int/